CLINICAL TRIAL: NCT05881525
Title: A Phase I/II Clinical Study of TC-N201 Injection for the Treatment of Advanced Solid Tumors With HLA-A2 Expression and Positive NY-ESO-1.
Brief Title: NY-ESO-1 TCR-T Cells for NY-ESO-1 Positive Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TCRCure Biopharma Ltd. (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TC-N201-ST
Record Dates: First submitted 2023-04-11; First posted 2023-05-31 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Interleukin-2; fludarabine; Cyclophosphamide; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- dose escalation (Experimental): This study uses the "3+3" dose escalation method. The initial dose is Dose 1, the maximum dose that patients can tolerate is determined as the phase II recommended dose (RPIID), and at least 6 patients are receiving RPIID treatment. If patients develop intolerance in Dose 1 (≥3 subjects with DLT), then the subsequent enrolled patients will receive Dose -1 infusion.
  Interventions:
  Biological: TCR-T cells Drug: IL-2 Drug: Fludarabine Drug: Cyclophosphamide Drug: Nab-Paclitaxel
  Interventions: Biological: TC-N201 cells; Drug: IL-2; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Nab-paclitaxel

INTERVENTIONS:
Biological: TC-N201 cells — T cells genetically engineered with a TCR targeting NY-ESO-1 (NY-ESO-1 TCR) that displays specific reactivity against HLA-A2+, NY-ESO-1+ target cells.
Drug: IL-2 — Following cell infusion, the patient receives intravenous IL-2. IL-2 improves the survival of TC-N201 cells after infusion.
Drug: Fludarabine — Part of the non-myeloablative lymphocyte-depleting preparative regimen.
Drug: Cyclophosphamide — Part of the non-myeloablative lymphocyte-depleting preparative regimen.
Drug: Nab-paclitaxel — Part of the non-myeloablative lymphocyte-depleting preparative regimen.

SUMMARY:
New York Esophageal Squamous Cell Carcinoma 1 (NY-ESO-1) is a cancer-testis antigen (CTA) which is expressed in various tumors. In TCR-T therapy, researchers take the blood of a certain patient, select T cells and insert genes into the cell that expressing a kind of protein that targeting NY-ESO-1. The genetically engineered cells are called NY-ESO-1 TCR-T cells. Then the engineered cells are re-infused to the cancer patients to cure the disease or prolong life.

DETAILED DESCRIPTION:
This is a single-center, open-label, Phase I clinical study of TCR-T cells for the treatment of the recurrent/metastatic solid tumors patients who had failed standard therapy.

Objective:

To evaluate the safety and efficacy of TCR-T cells for the treatment of advanced solid tumors.

Eligibility:

Adults aging 18-70 with advanced solid tumors

Design:

Patients will undergo screening tests, including imaging procedures, heart and lung tests, and lab tests.

Patients will have leukapheresis. Blood will be removed through a needle in the arm. A machine separates the white blood cells. The rest of the blood is returned through a needle in the other arm.

Engineered T cells will be re-infused into the patient. Patients will stay in hospital and be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Be able to understand and sign the Informed of Consent Document. Be willing to follow the procedure and protocol of the clinical trial;
* Age ≥ 18 years and ≤ 70 years;
* Expected survival time > 3 months;
* ECOG score 0-1;
* Metastatic or recurrent solid tumors confirmed by histopathology;
* Refractory to standard treatment evaluated by radiological assessment;
* Be able provide fresh or preserved tissue specimen;
* At least 1 measurable lesion (according to RECIST 1.1);
* NY-ESO-1 expression positive: Immunohistochemical staining positive cells ≥25% and positive staining intensity is "++" or above;
* HLA typing is HLA-A2 (excluding HLA-A*0203);
* Hematology should at least meet the following criteria:

  1. Absolute neutrophil count (ANC) ≥ 1.5× 109/L (±20%)；
  2. Platelet (PLT） ≥ 75× 109/L (±20%）；
  3. Hemoglobin (HGB) ≥ 90 g/L (±20%).
* Liver and kidney function are normal:

  1. Serum creatinine (Cr) ≤ 1.5 times of upper limit of normal (ULN) or creatine clearance ≥ 60 ml/min;
  2. Serum Alanine aminotransferase (ALT) or/and Aspartate aminotransferase (AST) ≤ 2.5 times of upper limit of normal;
  3. Total bilirubin (TBIL) ≤ 15 times of upper limit of normal.
* Blood coagulation function is normal: Prothrombin time (PT) ≤ 1.5 ULN, International Normalized Ratio (INR) ≤ 1.5 ULN, or Activated Partial Thromboplastin Time (APTT) ≤ 1.5 ULN;
* Echocardiogram results show: Left ventricular ejection fraction >45%;
* Women of childbearing potential should be ascetic or take contraception since the signing of ICF to 24 weeks or later after the last administration of drug Note: Women of childbearing age who have undergone surgical sterilization or who have already experienced menopause are considered to have no possibility of pregnancy.
* Before the TC-N201 injection was reconstituted, the toxic effects of standard treatment had already recovered, and the corresponding adverse events were judged by the researcher to not pose a safety risk;
* Catheter insertion is feasible and No White Blood Cells collection contraindications.

Exclusion Criteria:

* Under pregnancy or lactation, or positive based on blood pregnancy test;
* Severe allergic to related ingredients in the clinical trial;
* Received any other investigational treatment within 4 weeks before the first administration or enrolled in another clinical trial the same time;
* History of other known malignant tumors within the previous 5 years, including carcinoma in situ of the cervix, basal cell carcinoma of the skin, and carcinoma in situ of the prostate; Except for localized tumors that have been cured;
* Primary central nerve system (CNS) cancer, or subjects with CNS metastasis after localized treatment;
* Subjects with any active autoimmune disease, a history of autoimmune disease, or a history or syndrome requiring treatment with systemic steroids or immunosuppressive drugs;
* Immunodeficiency including HIV positive, harvested or natural immunodeficiency;
* Subjects with ≥ grade 3 thromboembolic events within 2 years or under thrombolysis treatment;
* Subjects with hereditary or acquired hemorrhagic disease;
* Have clinical cardiovascular disease or symptoms;
* Subjects with active infection: active infection requiring systemic anti-infective treatment (except topical antibiotics), fever caused by cancer could be enrolled according to the investigator's judgment;
* Subjects with active pulmonary tuberculosis infection detected by medical history or Computed Tomography (CT), or a history of active pulmonary tuberculosis infection within 1 year before enrollment, or a history of active pulmonary tuberculosis infection more than 1 year before enrollment but without regular treatment;
* Subjects with positive hepatitis B surface antigen or positive hepatitis B core antibody or positive hepatitis C virus antibody;
* Treponema pallidum antibody positive;
* Subjects received major surgery or under severe injury within 4 weeks before TC-N201 cell infusion;
* Subjects who received live vaccine or attenuated live vaccine 28 days before leukapheresis;
* Subjects who have drug addiction history, or alcoholism, drug users;
* Subjects who received cell therapy before enrollment，such as TCR-T，CAR-T and TIL;
* Subjects who have previously received treatment targeting NY-ESO-1;
* Subjects not suitable for the clinical trial according to investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity or Maximum Tolerated Dose (MTD) | Day 28 after the first TC-N201 infusion
  Dose Limiting Toxicity (DLT) is defined as patients with the adverse event (AE) or laboratory abnormality, and should be possibly related to TC-N201 cell therapy, and should be unrelated to the disease itself, disease progression, concomitant diseases or concomitant medication. MTD is defined as the highest dose at which ≤1 of 6 patients experienced a DLT or the highest dose level studied if DLTs are not observed at any of the dose levels.
Overall response rate | Day 0 - Day 730
  The efficacy of TC-N201 will be assessed by the objective response rate (ORR) evaluated according to RECIST 1.1 and iRECIST. ORR is described as patients assessed with partial response (PR) and complete response (CR).
Treatment-related adverse events as assessed by National Cancer Institute general terminology standard for adverse events (NCI CTCAE) v5.0 | Day 0 - Day 730
  The type, incidence and severity of adverse events include abnormal laboratory examination results with clinical significance after treatment, abnormal physical examination and blood examination results, bone marrow examination results, etc. Clinical and laboratory adverse events will be classified according to the CTCAE v5.0.

SECONDARY OUTCOMES:
Duration of response | Day 0 - Day 730
  The efficacy of TC-N201 will be assessed by duration of response (DOR). DOR refers to the length of time from the first appearance of a treatment response to the first occurrence of progressive disease or recurrence.
Progression free survival | Day 0 - Day 730
  The efficacy of TC-N201 will be assessed by progression free survival (PFS). PFS refers to the time from treatment to progressive disease or death for any reason.
Overall survival | Day 0 - Day 730
  The efficacy of TC-N201 will be assessed by overall survival (OS). OS refers to the time from treatment to death.
Maximum Persistence (Cmax) of TC-N201 | Day 0 - Day 730
  Blood samples were collected to measure persistence of infused TC-N201 using polymerase chain reaction of a vector specific sequence in deoxyribonucleic acid (DNA) extracted from peripheral blood mononuclear cell (PBMC).
Time to Maximum Persistence | Day 0 - Day 730
  Blood samples were collected to measure persistence of infused TC-N201 using polymerase chain reaction of a vector specific sequence in DNA extracted from PBMC.
Area Under the Plasma Concentration-time Curve From Zero to Day 28 (AUC [0-28]) | Day 28 after the first TC-N201 infusion
  Blood samples were collected to measure persistence of infused TC-N201 using polymerase chain reaction of a vector specific sequence in DNA extracted from PBMC.
Anti-PD-1 single chain antibody concentration | Day 0 - Day 730
  The pharmacodynamics of TC-N201 will be assessed by anti-PD-1 scFv.

CONTACTS AND LOCATIONS:
Overall Officials: ning Li, PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- TCRCure Biopharma Ltd., Chongqing, China

IPD SHARING:
Plan to Share IPD: No